CLINICAL TRIAL: NCT06457022
Title: Outcome Measures of Modified Constraint Induced Movement Therapy Versus Dual Task Training on Upper Extremity and Cognitive Functions in Patients With Hemiparesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahmed Alshimy (Other)
Responsible Party: Sponsor-Investigator, Ahmed Alshimy, Lecturer of Physical Therapy for Neurology and it's Surgery, AlRyada University for Science & Technology
Organization: AlRyada University for Science & Technology (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/005007
Record Dates: First submitted 2024-06-08; First posted 2024-06-13 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Hemiparesis
Keywords: Modified constraint induced movement therapy; Hemiparesis; Dual task training; Upper extremity; Cognitive functions
MeSH Terms: conditions — Paresis

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): Receiving modified constraint induced movement therapy , for 30 minutes , in addition to conventional physiotherapy program for the other 30 minutes.
  Interventions: Other: Modified Constraint Induced Movement therapy; Other: Conventional physiotherapy rehabilitation program
- Group B (Experimental): Receiving dual task training (Cognitive-Motor) for 30 minutes, in addition to conventional physiotherapy program for the other 30 minutes.
  Interventions: Other: Dual task training in the form of cognitive - motor task; Other: Conventional physiotherapy rehabilitation program
- Group C (Other): Receiving only conventional physiotherapy program for 60 minutes.
  Interventions: Other: Conventional physiotherapy rehabilitation program

INTERVENTIONS:
Other: Modified Constraint Induced Movement therapy — patient wears a restraint instrument in his unaffected hand, then applying massed practice to his affected upper extremity. The patient wears padded glove in his unaffected upper extremity for restraining the patient from using his unaffected upper extremity for about 3 hours per day including the treatment session and the home program. So, by this way the patient is reinforced to use his affected upper extremity during this period of time to achieve his activities of daily living. Finally, the total time, the patient spends it during the day wearing the glove should be recorded each day.
  Arms: Group A
Other: Dual task training in the form of cognitive - motor task — Verbal fluency: Ask the hemiparetic patient to title many words of specific type as fruits, vegetable or animals. Mental tracking: as the hemiparetic patient to subtract serial 3 between number 90 and 100.
  Arms: Group B
Other: Conventional physiotherapy rehabilitation program — Ultrasound on shoulder. Graduated active exercises for shoulder. Prolonged stretching for spastic muscles

SUMMARY:
All stroke patients were assessed via isokinetic dynamometer, Montreal cognitive assessment scale (MOCA) and Fugl Myer Upper extremity (FMUE) before and after the treatment program.

DETAILED DESCRIPTION:
The patients were classified randomly into three equal groups, Study group A (GA) receiving modified constraint induced movement therapy in addition to conventional physical therapy program, Study group B (GB) receiving dual task training in addition to conventional physical therapy program and control group C (GC) receiving only conventional physiotherapy program.

ELIGIBILITY:
Inclusion Criteria:

* Patients with age range between 55 and 65 years old.
* The patients were from both genders (males &females).
* Patients were of duration of illness between 6 and 12 months.
* The patients were scoring 1 &1+ on modified Ashworth scale (mild spasticity).
* The patients were of good ability to see and hear.
* Consent form was obtained from all participants to approve the study and follow the commands.
* All patients were scoring more than 26 on MMSE. All patients were medically stable.

Exclusion Criteria:

* patients with moderate and sever spasticity.
* patients with cognitive disorder due to other cause rather than spasticity.
* patients with unstable medical conditions.
* patients with previous or recurrent stroke.
* patients with respiratory problems.
* patients with shoulder dislocation or subluxation or frozen shoulder.
* patients with uncontrolled hypertension, diabetes mellitus, unstable angina or heart failure.

Ages: 55 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2024-06-10 (Actual); Primary Completion 2024-07-05 (Actual); Study Completion 2024-07-10 (Actual)

PRIMARY OUTCOMES:
Biodex isokinetic dynamometer | 4 weeks
  Used to assess muscle strength and function
Montreal cognitive assessment | 4 weeks
  a quick test that is used to examine mild cognitive impairment and early dementia.
Fugl Myer upper extremity | 4 weeks
  a scale used to measure the functional impairment of stroke

CONTACTS AND LOCATIONS:
Locations (1):
- Al Ryada University for Science and Technology, Sadat, Menoufia, Egypt

IPD SHARING:
Plan to Share IPD: No